CLINICAL TRIAL: NCT07311252
Title: Effectiveness of a Person-Centered Lifestyle Intervention in Mothers of Children With Autism Spectrum Disorder: A Randomized Controlled Trial With 6-Month Follow-Up
Brief Title: Effectiveness of a Person-Centered Lifestyle Intervention in Mothers of Children With Autism Spectrum Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ruya Gul Temel, PhD Candidate, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OT-ASD-KMYTM-2025
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder; Caregiver Burden; Quality of Life
MeSH Terms: conditions — Autism Spectrum Disorder; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm1 (Experimental): Person-Centered Lifestyle Intervention; Participants will receive a person-centered lifestyle intervention consisting of eight sessions delivered twice weekly over a one-month period.
  Interventions: Behavioral: Person-Centered Lifestyle Intervention
- arm2-control (No Intervention): Participants will continue their usual daily routines and will not receive the lifestyle intervention during the study period.

INTERVENTIONS:
Behavioral: Person-Centered Lifestyle Intervention — A structured person-centered lifestyle intervention delivered by occupational therapists, consisting of eight sessions over four weeks, focusing on individualized goal setting, occupational balance, stress management, and health-promoting routines.
  Arms: arm1

SUMMARY:
Mothers of children with autism spectrum disorder (ASD) experience substantial physical, emotional, and social strain due to the demands of continuous caregiving. These responsibilities often limit opportunities for health-promoting behaviors and contribute to elevated stress, fatigue, sleep disturbances, and reduced wellbeing. This study aims to evaluate an intervention designed to support the health and wellbeing of mothers who serve as primary caregivers of children with ASD. The intervention focuses on enhancing stress-management skills, improving participation in meaningful daily activities, and promoting balanced health behaviors through structured psychoeducational and occupation-based strategies. The goal of the trial is to determine whether a holistic, individualized, and occupation-centered approach delivered by occupational therapists can improve maternal wellbeing and support sustainable engagement in health-promoting routines.

DETAILED DESCRIPTION:
Caregivers provide extensive support to individuals with special needs across the lifespan by assisting with daily living activities and health-related needs. In many societies, caregiving is primarily assumed as a family responsibility, and women, particularly mothers, most often undertake the primary caregiving role for children with special needs. Mothers of children with autism spectrum disorder frequently devote substantial time and energy to caregiving tasks and to facilitating their children's participation in daily life, which may limit opportunities for self-care, health-promoting activities, rest, and access to healthcare services.

Autism spectrum disorder is a highly heterogeneous condition that requires long-term and multifaceted support across educational, health, and social domains. The continuous caregiving demands associated with autism spectrum disorder place mothers at increased risk for physical strain, psychological distress, reduced quality of life, and disruptions in daily routines. Caregiving is a subjective experience, and the needs and expectations of caregivers of children differ from those caring for adults, highlighting the importance of individualized and context-sensitive interventions.

Most existing interventions for caregivers focus primarily on improving parenting skills or child outcomes, while fewer programs directly target caregiver health and wellbeing. Evidence suggests that interventions incorporating cognitive, behavioral, and educational components may support stress management, problem-solving skills, and healthy lifestyle behaviors. However, no single intervention approach adequately addresses the complex and individualized needs of caregiving mothers.

This study is designed as a randomized controlled trial with a six-month follow-up period to examine the effectiveness of a person-centered lifestyle intervention for mothers who are primary caregivers of children diagnosed with autism spectrum disorder. Participants will be randomly assigned to an intervention group or a control group using a computer-assisted randomization process. The intervention consists of eight sessions delivered twice weekly over one month and focuses on individualized goal setting, occupational balance, health-promoting routines, stress management strategies, and meaningful participation in daily activities. The control group will continue their usual daily routines without receiving the intervention during the study period.

Outcomes related to occupational performance and satisfaction, caregiver burden, psychological status, and health-related quality of life will be assessed at baseline, immediately following the intervention, and at six months to evaluate short-term and sustained effects of the intervention. The study adopts a holistic, biopsychosocial, and person-centered approach consistent with occupational therapy practice, with the aim of informing future caregiver-focused interventions in pediatric rehabilitation.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* Mother of a child with a medically confirmed diagnosis of autism spectrum disorder
* Primary caregiver and living with the child
* Age 18 years or older
* Ability to participate in all intervention sessions and assessments

Exclusion Criteria:

* Pregnancy or postpartum period
* Having more than one child with a disability
* Participation in a similar lifestyle or caregiver intervention program within the past year
* Presence of a diagnosed severe physical, mental, or psychiatric condition that would interfere with participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Occupational Performance and Satisfaction Occupational Performance and Satisfaction | Baseline, immediately post-intervention (1 month), and 6 months follow-up
  Occupational performance and satisfaction will be assessed using the Canadian Occupational Performance Measure. Participants identify meaningful daily activities and rate their performance and satisfaction with performance on a 10-point scale. Higher scores indicate better occupational performance and greater satisfaction.

SECONDARY OUTCOMES:
Caregiver Burden | Baseline, immediately post-intervention (1 month), and 6 months follow-up
  Caregiver burden will be evaluated using the Zarit Caregiver Burden Interview, which assesses the perceived impact of caregiving responsibilities on emotional, social, and physical wellbeing. Higher scores indicate greater caregiver burden.
Psychological Status | Baseline, immediately post-intervention (1 month), and 6 months follow-up
  Psychological status will be assessed using the Depression Anxiety Stress Scale, which measures symptoms related to depression, anxiety, and stress. Higher scores reflect greater psychological distress.
Health-Related Quality of Life | Baseline, immediately post-intervention (1 month), and 6 months follow-up
  Health-related quality of life will be assessed using the Nottingham Health Profile, which evaluates perceived health problems across physical, emotional, and social domains. Higher scores indicate poorer perceived health status.